CLINICAL TRIAL: NCT03219697
Title: Preventing and Addressing At-obesity-Risk Early Years INtervention with Home Visits in Toronto (PARENT): a Pragmatic RCT
Acronym: PARENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); The Physicians' Services Incorporated Foundation (Other); Ontario Child Health Support Unit (Unknown)
Responsible Party: Principal Investigator, Catherine Birken, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1000054998
Record Dates: First submitted 2017-06-27; First posted 2017-07-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Child Obesity
Keywords: Childhood obesity prevention;
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parenting education program (Experimental): 8 weeks of group parenting education sessions followed by two optional booster sessions.
  2 public health nurse home/virtual visits and 4 coaching calls over a period of 6 months.
  Interventions: Behavioral: Parenting education program
- Control (No Intervention): Receive regular health care

INTERVENTIONS:
Behavioral: Parenting education program — 8-week parent/caregiver education program, followed by two booster sessions. You and/or your partner will attend weekly parenting sessions which will take place either at the office of your child's primary care provider or virtually. Our Toronto Public Health Nurse, will arrange 2 home visits/virtual visits with you and your family along with 4 coaching calls during the 6 months. This first home visit will include learning more about your routines at home, and what is available in your neighbourhood. The home visits will focus on helping to apply the messages and skills from the group sessions for your family, and making connections in your community that you find helpful such as recreational or nutrition programs or other supports for your family.
  Arms: Parenting education program

SUMMARY:
The PARENT Trial aims to determine if the Parents Together program consisting of parent workshops, home visits and coaching calls, will result in better health outcomes for children. The program which is facilitated by a Public Health Nurse seeks to encourage healthy lifestyle, help build strong family relationships, and promote child mental health.

DETAILED DESCRIPTION:
This study will determine whether a primary care based intervention that combines group based parenting skills training and public health nurse home visits with a focus on healthy nutrition, activity and sleep, compared to regular health care will lead to improved weight status in 18 months- 4 year old children.

Healthy children at risk for obesity will be identified through primary care practices participating in TARGet Kids!. Families who participate in this study will be randomly assigned (having an equal chance of being in either group) to one of the two study groups that will run for 6-months:

Group A: Receive 8 weeks of group parenting education sessions, 2 additional group sessions, with 2-4 public health nurse home/virtual visits Group B: Receive regular health care

ELIGIBILITY:
Inclusion Criteria:

* Children at risk for childhood obesity (meeting any of the risk factors below):
* birth weight greater than 3500g
* weight gain in first year of life (crossing of at least 1 percentile line of weight for age or weight for length percentile)
* maternal or paternal obesity,
* gestational smoking at birth
* low median household self-reported income
* availability of at least one caregiver to participate in trial

Exclusion Criteria:

* Young children with Prader-Willi syndrome or severe developmental delays
* obesity or severe obesity (defined as zBMI >2 for all ages)
* families not fluent in English
* children with a sibling already enrolled in the study
* families who reside beyond the Toronto Public Health catchment areas

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
zBMI | at 6 months and 12 months post-randomization
  Measure the difference in age and sex-standardized BMI z-score (zBMI)

SECONDARY OUTCOMES:
Mental health | at 6 months and 12 months post-randomization
  Assess mental health by Strengths and Difficulties Questionnaire
Eating behaviour and dietary intake | at 6 months and 12 months post-randomization
  Assess eating behaviour and dietary intake using the Nutrition Screening Tool for Every Preschooler (NutriSTEP)
ZBMI | at 6 months and 12 months post-randomization
  Measure the difference in age and sex-standardized BMI z-score (zBMI)
Physical Activity, Sedentary Time, Sleep Duration | at 6 months and 12 months post-randomization
  Parent reported measures of physical activity, sedentary time, and sleep duration (based on the Canadian Community Health Survey),
Physical Activity | At 12 months post-randomization
  Direct measures of physical activity using accelerometry
Psychosocial Health | at 6 months and 12 months post-randomization
  family psychosocial health (using the Parental Stress Index)
Maternal Mental Health | at 6 months and 12 months post-randomization
  maternal mental health (Depression Anxiety Stress Scale and Patient Health Questionnaire)
Parenting | at 6 months and 12 months post-randomization
  Parenting (using the Parenting Scale)
sociodemographic, maternal and child characteristics | at 6 months and 12 months post-randomization
  parent self-reported income, maternal education, ethnicity, immigration status, and marital status, questions about parents health, exposures during pregnancy, family medical history - captured by the Nutrition and Health Questionnaire (NHQ).
Waist circumference | 6 and 12 months post randomization
  measured waist circumference using a tape measure
blood pressure | 6 and 12 months post-randomization
  measurement of diastolic and systolic blood pressure in children 3 years of age and older
laboratory measures of cardiometabolic risk | At 12 months post-randomization
  laboratory measures of cardiometabolic risk (cholesterol, insulin, glucose), iron and vitamin D status
Feasibility of intervention | at 12 months post randomization
  1. feasibility of study design (i.e., recruitment, outcome assessment)
  2. feasibility of intervention (i.e., intervention fidelity)
  3. acceptability of study design (i.e., randomization),
  4. acceptability of intervention (i.e., attendance, parent satisfaction).
Cost effectiveness analysis | at 12 months post-randomization
  to determine the incremental costs of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Catherine S Birken, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - St Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rae S, Maguire J, Aglipay M, Barwick M, Danavan K, Haines J, Jenkins J, Klaassen M, Moretti ME, Ong F, Persaud N, Porepa M, Straus S, Tavares E, Willan A, Birken C. Randomized controlled trial evaluating a virtual parenting intervention for young children at risk of obesity: study protocol for Parenting Addressing Early Years Intervention with Coaching Visits in Toronto (PARENT) trial. Trials. 2023 Jan 4;24(1):8. doi: 10.1186/s13063-022-06947-w. PMID 36600302